CLINICAL TRIAL: NCT02820467
Title: Study of Parameters of Infracyanine Angiography as Diagnostic Tool of Critical Limb Ischemia
Brief Title: Use of Indocyanine Green Angiography in Critical Limb Ischemia
Acronym: FLUORESCENCE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC15.212
Record Dates: First submitted 2016-06-10; First posted 2016-07-01 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Indocyanine; Angiography; Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Ischemia | interventions — Fluorescein Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patients with suspicion of CLI (Experimental): patients presenting with peripheral artery disease and suspicion of critical limb ischemia as assessed by TASK II consensus 30 patients will be enrolled and will benefit of measures of TcPO2, too systolic blood pressure and skin perfusion pressure and in the same time angiography with fluorescence (Indocyanine grey 0.05 mg/kg by intravenous injection
  Interventions: Device: fluorescence angiography

INTERVENTIONS:
Device: fluorescence angiography — Injection of indocyanine grey in an antecubital vein at the posology of 0.05 mg/kg

SUMMARY:
Investigators conduct a monocentric pilot study with the objective to determine the hemodynamic parameter of fluorescence angiography (slope, amplitude, saturation time ) best correlated with toe pressure in patients with suspicion of critical limb ischemia.

DETAILED DESCRIPTION:
Critical limb ischemia, defined as the presence of chronic ischemic rest pain, ulcers or gangrene attributable to objectively proven arterial occlusive disease, is associated with the appalling prospect that approximately 30% will lose their leg and 25% will die at one year. Despite the progress of therapeutics these statistics haven't changed. Critical limb ischemia is a clinical diagnosis but should be supported by objective tests. None of theses tests (toe blood pressure (TBP), transcutaneous oxygen pressure (TcPO2) and skin perfusion pressure (SPP)) have proven to be enough specific or sensitive, more so they are time consuming, can be subject to several artifacts and may be in some cases discordant making diagnosis difficult. Fluorescence angiography has long been used in ophthalmology for the evaluation of the microcirculation of the retina. Infracyanine remains within the intravascular space allowing the visualization of the vasculature to a depth of 10 mm. With the Fluobeam system, images to a maximal width of 20 cm can be obtained therefore allowing the evaluation of the tissue perfusion of the entire foot.

Method: Fluorescence angiography is performed in the laboratory in the same time as TCPO2, TP and SPP. Infracyanine is injected in an antecubital vein and visualization and signal acquisition carried out using a specific camera device (Fluoptic SAS, France) producing the time course of hemodynamic parameters (slope, amplitude, saturation time).

30patients will be evaluated with correlation between data obtained by fluorescence angiography and too blood pressure

ELIGIBILITY:
Inclusion Criteria:

* patients with peripheral artery disease and suspicion of critical limb ischemia

Exclusion Criteria:

* pregnant women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Correlation of parameters of fluorescence on time intensity curve ( saturation time (s) with toe pressure (mm hg) assessed by laser doppler | instantaneous, at the time the exam is performed
Correlation of parameters of fluorescence on time intensity curve ( amplitude (UA) with toe pressure (mm hg) assessed by laser doppler | instantaneous, at the time the exam is performed
Correlation of parameters of fluorescence on time intensity curve ( slope) with toe pressure (mm hg) assessed by laser doppler | instantaneous, at the time the exam is performed

SECONDARY OUTCOMES:
Correlation of parameters of fluorescence on time intensity curve ( saturation time (s) with transcutaneous cutaneous pressure of oxygen (mm Hg) | instantaneous, at the time the exam is performed
Correlation of parameters of fluorescence on time intensity curve ( amplitude (UA) with transcutaneous cutaneous pressure of oxygen (mm Hg) | instantaneous, at the time the exam is performed
Correlation of parameters of fluorescence on time intensity curve (slope) with transcutaneous cutaneous pressure of oxygen (mm Hg) | instantaneous, at the time the exam is performed

CONTACTS AND LOCATIONS:
Overall Officials: christophe seinturier, MD, Principal Investigator — CHU Grenoble france
Locations (1):
- CHU grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Becker F, Robert-Ebadi H, Ricco JB, Setacci C, Cao P, de Donato G, Eckstein HH, De Rango P, Diehm N, Schmidli J, Teraa M, Moll FL, Dick F, Davies AH, Lepantalo M, Apelqvist J. Chapter I: Definitions, epidemiology, clinical presentation and prognosis. Eur J Vasc Endovasc Surg. 2011 Dec;42 Suppl 2:S4-12. doi: 10.1016/S1078-5884(11)60009-9. PMID 22172472
- [Background] Bloch C, Richard JL. [Risk factors for atherosclerotic diseases in the Prospective Parisian Study I. Comparison with foreign studies]. Rev Epidemiol Sante Publique. 1985;33(2):108-20. French. PMID 3898252
- [Background] Braun JD, Trinidad-Hernandez M, Perry D, Armstrong DG, Mills JL Sr. Early quantitative evaluation of indocyanine green angiography in patients with critical limb ischemia. J Vasc Surg. 2013 May;57(5):1213-8. doi: 10.1016/j.jvs.2012.10.113. Epub 2013 Jan 24. PMID 23352361
- [Background] Chung J, Modrall JG, Valentine RJ. The need for improved risk stratification in chronic critical limb ischemia. J Vasc Surg. 2014 Dec;60(6):1677-85. doi: 10.1016/j.jvs.2014.07.104. Epub 2014 Sep 8. PMID 25214365
- [Background] Ciardella AP, Prall FR, Borodoker N, Cunningham ET Jr. Imaging techniques for posterior uveitis. Curr Opin Ophthalmol. 2004 Dec;15(6):519-30. doi: 10.1097/01.icu.0000144386.05116.c5. PMID 15523198
- [Background] Constans J, Bura-Riviere A. [Lower limb occlusive arterial disease: Diagnosis problems in 2014]. Presse Med. 2014 Jul-Aug;43(7-8):823-6. doi: 10.1016/j.lpm.2014.03.013. Epub 2014 Jun 2. French. PMID 24890636
- [Background] Cull DL, Manos G, Hartley MC, Taylor SM, Langan EM, Eidt JF, Johnson BL. An early validation of the Society for Vascular Surgery lower extremity threatened limb classification system. J Vasc Surg. 2014 Dec;60(6):1535-41. doi: 10.1016/j.jvs.2014.08.107. Epub 2014 Oct 3. PMID 25282695
- [Background] Elsayed S, Clavijo LC. Critical limb ischemia. Cardiol Clin. 2015 Feb;33(1):37-47. doi: 10.1016/j.ccl.2014.09.008. PMID 25439329
- [Background] Terasaki H, Inoue Y, Sugano N, Jibiki M, Kudo T, Lepantalo M, Venermo M. A quantitative method for evaluating local perfusion using indocyanine green fluorescence imaging. Ann Vasc Surg. 2013 Nov;27(8):1154-61. doi: 10.1016/j.avsg.2013.02.011. Epub 2013 Aug 20. PMID 23972435
- [Background] Igari K, Kudo T, Toyofuku T, Jibiki M, Inoue Y, Kawano T. Quantitative evaluation of the outcomes of revascularization procedures for peripheral arterial disease using indocyanine green angiography. Eur J Vasc Endovasc Surg. 2013 Oct;46(4):460-5. doi: 10.1016/j.ejvs.2013.07.016. Epub 2013 Aug 21. PMID 23973274
- [Background] Kang Y, Lee J, Kwon K, Choi C. Application of novel dynamic optical imaging for evaluation of peripheral tissue perfusion. Int J Cardiol. 2010 Dec 3;145(3):e99-101. doi: 10.1016/j.ijcard.2008.12.166. Epub 2009 Feb 23. PMID 19230993
- [Background] Kang Y, Lee J, Kwon K, Choi C. Dynamic fluorescence imaging of indocyanine green for reliable and sensitive diagnosis of peripheral vascular insufficiency. Microvasc Res. 2010 Dec;80(3):552-5. doi: 10.1016/j.mvr.2010.07.004. Epub 2010 Jul 15. PMID 20637783
- [Background] Kannel WB, McGee DL. Update on some epidemiologic features of intermittent claudication: the Framingham Study. J Am Geriatr Soc. 1985 Jan;33(1):13-8. doi: 10.1111/j.1532-5415.1985.tb02853.x. PMID 3965550
- [Background] Labs KH, Dormandy JA, Jaeger KA, Stuerzebecher C, Hiatt WR. Trans-atlantic conference on clinical trial guidelines in PAOD (Peripheral arterial occlusive disease) clinical trial methodology. Eur J Vasc Endovasc Surg. 1999 Sep;18(3):253-65. doi: 10.1053/ejvs.1999.0931. No abstract available. PMID 10480800
- [Background] Levesque E, Hoti E, Azoulay D, Adam R, Samuel D, Castaing D, Saliba F. Non-invasive ICG-clearance: a useful tool for the management of hepatic artery thrombosis following liver transplantation. Clin Transplant. 2011 Mar-Apr;25(2):297-301. doi: 10.1111/j.1399-0012.2010.01252.x. PMID 20412097
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Pestana IA, Coan B, Erdmann D, Marcus J, Levin LS, Zenn MR. Early experience with fluorescent angiography in free-tissue transfer reconstruction. Plast Reconstr Surg. 2009 Apr;123(4):1239-1244. doi: 10.1097/PRS.0b013e31819e67c1. PMID 19337092
- [Background] Rashid H, Slim H, Zayed H, Huang DY, Wilkins CJ, Evans DR, Sidhu PS, Edmonds M. The impact of arterial pedal arch quality and angiosome revascularization on foot tissue loss healing and infrapopliteal bypass outcome. J Vasc Surg. 2013 May;57(5):1219-26. doi: 10.1016/j.jvs.2012.10.129. Epub 2013 Mar 21. PMID 23523278
- [Background] Schaafsma BE, Mieog JS, Hutteman M, van der Vorst JR, Kuppen PJ, Lowik CW, Frangioni JV, van de Velde CJ, Vahrmeijer AL. The clinical use of indocyanine green as a near-infrared fluorescent contrast agent for image-guided oncologic surgery. J Surg Oncol. 2011 Sep 1;104(3):323-32. doi: 10.1002/jso.21943. Epub 2011 Apr 14. PMID 21495033
- [Background] Yamada T, Ohta T, Ishibashi H, Sugimoto I, Iwata H, Takahashi M, Kawanishi J. Clinical reliability and utility of skin perfusion pressure measurement in ischemic limbs--comparison with other noninvasive diagnostic methods. J Vasc Surg. 2008 Feb;47(2):318-23. doi: 10.1016/j.jvs.2007.10.045. PMID 18241755
- [Background] Zimmermann A, Roenneberg C, Reeps C, Wendorff H, Holzbach T, Eckstein HH. The determination of tissue perfusion and collateralization in peripheral arterial disease with indocyanine green fluorescence angiography. Clin Hemorheol Microcirc. 2012;50(3):157-66. doi: 10.3233/CH-2011-1408. PMID 22240349